CLINICAL TRIAL: NCT03552211
Title: Evaluation of the Incidence of Relapses in Patients With Biotin-treated Progressive Multiple Sclerosis
Acronym: IPBio-SeP
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: OFSEP (Observatoire Français de la Sclérose en Plaques) (Unknown); SFSEP (Société Francophone de la Sclérose en Plaques) (Unknown); MedDay Pharmaceuticals SA (Industry)
Responsible Party: Sponsor
Other Study IDs: CHU-388
Record Dates: First submitted 2018-04-25; First posted 2018-06-11 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-05

CONDITIONS: Progressive Multiple Sclerosis
Keywords: Multiple Sclerosis; Progressive Multiple Sclerosis; Biotin; Relapse
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis; Recurrence | interventions — Biotin; Propensity Score

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients treated with biotin: This is a national, academic, observational and retrospective study comparing one group of progressive MS patients with high dose biotin to another group without this treatment using a propensity score, in intention to treat
  Interventions: Drug: biotin
- Control patients: This is a national, academic, observational and retrospective study comparing one group of progressive MS patients with high dose biotin to another group without this treatment using a propensity score, in intention to treat
  Interventions: Other: propensity score

INTERVENTIONS:
Drug: biotin — This is a national, academic, observational and retrospective study comparing one group of progressive MS patients with high dose biotin to another group without this treatment using a propensity score, in intention to treat.
  Groups: Patients treated with biotin
Other: propensity score — This is a national, academic, observational and retrospective study comparing one group of progressive MS patients with high dose biotin to another group without this treatment using a propensity score, in intention to treat.
  Groups: Control patients

SUMMARY:
Background: High dose biotin is a therapeutic option for French progressive Multiple Sclerosis (MS) patients, without relapse for at least one year, since June 1, 2016. Despite the inflammatory activity of progressive forms of MS is known to be low, several publications mentioned clinical and/or radiological activity for biotin-treated patients.

Objectives:

1. To determine if high dose biotin increase the clinical inflammatory activity of patients with a progressive form of MS.
2. To compare the clinical characteristics of the relapses that occurred with biotin or not.
3. To describe the characteristics of the patients with a clinical inflammatory activity with biotin.

Methods: This is a national, academic, observational and retrospective study comparing one group of progressive MS patients with high dose biotin to another group without this treatment using a propensity score, in intention to treat. The main judgment criterion is the annualized relapse rate (ARR) from the beginning of the biotin to the last evaluation available before the data extraction. A Student's t test will be used. A negative binomial modelling with relapses counting over a period of exposure and taking into account the inter and intra center variability will be used. The statistical tests will be adapted to the nature of the variables concerning the secondary judgment criteria.

Expected results: This French national study will provide a better knowledge of the inflammatory activity of the progressive forms of MS treated with high dose biotin. If an increased clinical inflammatory activity is highlighted with biotin a prospective study will be necessary to confirm the result before a specific information of the scientific community and the patients about this risk or even an amendment of prescription rules in order to secure the use of the product. On the contrary, the absence of increased risk of clinical inflammatory activity with biotin would help to reassure the prescriber and the patient about the innocuity of the treatment.

DETAILED DESCRIPTION:
Investigators are going to recruit retrospectively all the patients treated with biotin since the product is available in France, in all French MS centers that agree to participate (maximum 30). They are going to collect through medical records, demographic data (as age, gender, MS center localization), but also data about the disease (as MS duration, primary progressive or secondary progressive MS), data about disability (with several Expanded Disability Status Scale -EDSS- scores at different time points) and data about treatments (as duration of biotin, existence of other concomitant disease-modifying therapy). For comparison, a control group without biotin is going also to be recruited from the European Database for Multiple Sclerosis (EDMUS). The same data as described above are going to be collected for the controls.

ELIGIBILITY:
Inclusion Criteria:

* For the patients treated with biotin :
* progressive form of MS (primary or secondary)
* age between 18 and 80 years
* Expanded Disability Status Scale (EDSS) between 3 and 7.5 at the beginning of biotin
* treatment with biotin 300 mg per day at least one time, ongoing or stopped
* no relapse in the year preceding biotin introduction
* follow-up in an MS expert center
* For the controls :
* progressive form of MS (primary or secondary)
* age between 18 and 80 years
* Expanded Disability Status Scale (EDSS) between 3 and 7.5 at the baseline
* EDMUS data base fulfilled at least three times during the two previous years
* no relapse in the year preceding the baseline
* follow-up in an MS expert center

Exclusion Criteria:

* For all participants :
* other disease modifying therapy (DMT) than interferon, methotrexate, mycophenolate mofetil, azathioprine, rituximab, ocrelizumab
* For the controls :
* treatment with biotin actually or in the past
* follow-up in an MS expert center who do not provide exhaustive information about biotin

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Progressive forms of Multiple Sclerosis
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2018-05-30 (Estimated); Primary Completion 2019-02-01 (Estimated); Study Completion 2019-04-30 (Estimated)

PRIMARY OUTCOMES:
Relapses with biotin | at day 1 (through study completion, an average of 1 year)
  To determine if high dose biotin increases the clinical inflammatory activity of patients with a progressive form of MS using the annualized relapse rate (ARR) comparing to a control group

SECONDARY OUTCOMES:
Clinical characteristics of the relapses with biotin | at day 1 (through study completion, an average of 1 year)
  To compare the clinical characteristics of the relapses that occurred with biotin or not.
Characteristics of patients with relapse with biotin | at day 1 (through study completion, an average of 1 year)
  To describe the characteristics of the patients with a clinical inflammatory activity with biotin

CONTACTS AND LOCATIONS:
Overall Officials: Pierre CLAVELOU, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-FERRAND, Clermont-Ferrand, France